CLINICAL TRIAL: NCT04433871
Title: National SFCE Cohort of SARS-CoV-2 Infections (COVID-19) in Pediatric Oncology and Hematology
Brief Title: COVID-19 in Pediatric Oncology and Hematology Centers in France
Acronym: PEDONCOVID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 20-065
Record Dates: First submitted 2020-04-24; First posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-04

CONDITIONS: Covid-19; Cancer
Keywords: child
MeSH Terms: conditions — COVID-19; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention, observational — No intervention, observational

SUMMARY:
Since the description of the first cases of infection in December 2019 in the Hubei province in China, a new coronavirus, called SARS-CoV-2 (severe acute respiratory syndrome coronavirus 2), emerged and caused a pandemic. This new virus is responsible for an infectious disease with respiratory and potent severe symptoms, called COVID-19 (coronavirus disease 2019). The first data concerned essentially the adult population and gave a clinical description of the disease. However, data is missing in the pediatric population. The first published studies indicate that children seem to have a lower risk to get a severe form of COVID-19. Except the case of a child with leukemia recently described with the diagnosis of COVID-19, there is currently no data about pediatric patients with an oncology history or under chemotherapeutic drugs. Cancers are rare among children and is estimated to concern about 1700 new cases in a year in France. Malignant tumor or its treatment can affect self-immunity, which could favor SARS-CoV-2 infection or its aggravation. Thus, the investigators propose in this study to collect data about French children with a cancer and diagnosed with COVID-19.The analysis of the collected data will refine clinical characteristics of SARS-CoV-2 infection in this population. It will be critical for elaborating recommendations for the management of COVID-19 in children with cancer.

DETAILED DESCRIPTION:
Since the description of the first cases in December 2019, the world is facing the emergence of a new coronavirus called "severe acute respiratory syndrome coronavirus 2" (SARS-CoV-2), which is responsible for an infectious disease mainly with respiratory manifestation and potently severe or even lethal, named coronavirus disease 2019 (COVID-19) (N. Zhu et al. 2020; Huang et al. 2020). The global spread of this virus led to the development of an unprecedented pandemic with an huge impact on public health and from a social and economic point of view (Ayittey et al. 2020).

First published data mainly concerned the adult population with a detailed COVID-19 clinical description. Few data are available in children. However, the first studies suggest that children may be at a lower risk than adults of developing a severe form of COVID-19 (Guan et al. 2020; Lu et al. 2020; Sinha et al. 2020). Neonatal presentation may be more severe (H. Zhu et al. 2020). Children seem to present with similar symptoms compared with adults but often with a milder form (Cao et al. 2020). Radiological findings also appear to be similar to those in adults (Liu et al. 2020; Xia et al. 2020). Children may be asymptomatic and may participate in the spread of SARS-CoV-2 (Lu et al. 2020; Chan et al. 2020). Nevertheless, severe COVID-19 forms were described in children, even if deaths remain extremely rare (Sun et al. 2020; Lu et al. 2020). Among the previous described severe forms, one of the patient dependent on mechanic ventilation had acute lymphoblastic leukemia (Sun et al. 2020). The publication of Lu et al. probably refers to this patient and it appears that this patient was receiving a maintenance treatment (Lu et al. 2020). This patient presented a co-infection with influenza virus, which probably explained his aggravation (Sun et al. 2020).

To describe COVID-19 presentation in children, adolescent and young adults, this study will include all patients with the following criteria:

- Patient followed-up in any French pediatric oncology and hematology center for a cancer or a benign tumor treated with chemotherapy, radiotherapy or a targeted therapy and with an oncologic treatment ongoing or terminated within the last 6 months, or with an hematopoietic stem cell transplantation history with an immunosuppressive treatment ongoing or terminated within the last 6 months, or a CAR-T cell therapy history

AND

- PCR or serologically-confirmed SARS-CoV-2 infection

OR

-Clinical and radiological diagnosis of SARS-CoV-2 infection with the following criteria : At least two of the following signs (three if no history of contact with an individual with a confirmed COVID-19): fever, cough, loss of smell, loss of taste, myalgia, chest pain, breath shortness, rhinorrhea, acute respiratory signs, diarrhea, headache, recent lethargy, skin rash.

AND

- At least one abnormality compatible with COVID-19 on a chest computed tomography scan.

In all included patients, the following informations will be retrieved from their medical record :

* socio-demographic and anthropometric data: age, sex, weight, height...
* cancer history: type of cancer, severity, ongoing or 30-days past oncologic treatment, significant oncologic treatment with potent impact on COVID-19 evolution (lung surgery, lung radiotherapy...)
* clinical symptoms at initial stage, at 10-15, 15-20, 20-30 days of evolution
* biological signs at initial stage, at 10-15, 15-20, 20-30 days of evolution
* radiological signs at initial stage and on the following exams
* COVID-19 management data: oxygen, antiviral agents, antibiotics...
* Evolutive data: resolution/aggravation of infection, potent sequelae...

ELIGIBILITY:
Inclusion Criteria:

* Children and parents or adult patient informed AND
* Patient followed-up in a French SFCE pediatric oncology and/or hematology center AND
* Patient followed-up for a cancer or a benign tumor treated with chemotherapy, radiotherapy or targeted therapy and an oncologic treatment ongoing or terminated less than 6 months ago, or patient with an history of hematopoietic stem cells transplantation with immunosuppressive treatment ongoing or terminated less than 6 month ago, or patient with history of CAR-T cell therapy AND
* SARS-CoV-2 infection confirmed by PCR or IgM positivity OR
* Compatible diagnosis of SARS-CoV-2 infection without biological confirmation if: 1- presence of at least two of the following clinical signs if any contact with a COVID+ subject or three of the following clinical signs in case of no such contact: fever, cough, taste or smell abnormality, myalgia, rhinorrhea, diarrhea, respiratory acute signs, recent fatigue, rash, chest pain. AND
* At least one chest CT-scan abnormality compatible with COVID-19

Exclusion Criteria:

* opposition of the patient or of the parents

Ages: 1 Month to 30 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children or young adult with a recent oncologic history diagnosed with COVID-19.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-04-27 (Actual); Primary Completion 2022-04-27 (Estimated); Study Completion 2023-04-27 (Estimated)

PRIMARY OUTCOMES:
Oncologic data | through study completion, an average of 1 year
  Type of cancer and/or underlying pathologies, oncologic treatments administrated before COVID-19 diagnosis.
COVID-19 diagnosis | through study completion, an average of 1 year
  Date of COVID-19 diagnosis, method of diagnosis (PCR and/or clinical signs and/or serology)
Clinical signs | through study completion, an average of 1 year
  Description of clinical signs at initial phase, days 7-10, days 15-20 and days 25-30
Biological signs | through study completion, an average of 1 year
  Description of biological signs at initial phase, days 7-10, days 15-20 and days 25-30
Radiological signs | through study completion, an average of 1 year
  chest X-rays and/or CT-scan description if performed
COVID-19 management | through study completion, an average of 1 year
  Management in hospital or at home, use of specific drugs against SARS-CoV2, oxygen required or not, other drugs administrated to manage infection complications.
Potent COVID-19 sequelae | through study completion, an average of 1 year
  type of sequelae if any

CONTACTS AND LOCATIONS:
Overall Officials: Jérémie Rouger-Gaudichon, MD, PhD, Principal Investigator — University Hospital of Caen
Locations (1):
- Jérémie Rouger-Gaudichon, Caen, France

IPD SHARING:
Plan to Share IPD: Undecided